CLINICAL TRIAL: NCT04352738
Title: Deciphering the Role of the Liver in Glucose Homeostasis Using Metabolic Imaging
Brief Title: Role of the Liver in Glucose Homeostasis Using Metabolic Imaging
Acronym: LEMON
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Principal Investigator, Lia Bally, Professor, Insel Gruppe AG, University Hospital Bern
Other Study IDs: LEMON
Record Dates: First submitted 2020-04-15; First posted 2020-04-20 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Type 1 Diabetes; Bariatric Surgery Candidate
Keywords: Hepatic glucose metabolism; Deuterium metabolic imaging; Insulin and glucose kinetics; Metabolic imaging
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy adults (group I)
  Interventions: Diagnostic Test: Multiparametric, multinuclear MR (DMI/ 13C-MRS/ GlycoCEST/GlycoNOE)
- Adults with type 1 diabetes (group II): * T1D for ≥2 years or evidence of undetectable C-peptide (<100pmol/l with concomitant plasma glucose≥4.0mmol/l).
  * HbA1c≤8.0mmol/l (64mmol/mol).
  Interventions: Diagnostic Test: Multiparametric, multinuclear MR (DMI/ 13C-MRS/ GlycoCEST/GlycoNOE)
- Adults after bariatric surgery (group III): * Female.
  * Bariatric surgery (Roux-en-Y gastric bypass or sleeve gastrectomy) ≥1 year ago.
  * Lack of a history of diabetes or pre-diabetes (HbA1c≤5.6% in the absence of anaemia).
  Interventions: Diagnostic Test: Multiparametric, multinuclear MR (DMI/ 13C-MRS/ GlycoCEST/GlycoNOE)

INTERVENTIONS:
Diagnostic Test: Multiparametric, multinuclear MR (DMI/ 13C-MRS/ GlycoCEST/GlycoNOE) — Magnetic resonance scanning for 150 minutes involving ingestion of 60g of 6,6, 2H2-glucose diluted in 200ml of tap water. Frequent blood samples will be drawn for measurements of plasma glucose, insulin, C-peptide and glucagon

SUMMARY:
The primary objective of this study is to assess hepatic glucose uptake using non-invasive metabolic imaging in three different populations that differ in terms of insulin and glucose kinetics. Between-group comparison will address the following two hypotheses:

i) Hepatic glucose uptake will be lower in participants with type 1 diabetes compared with matched controls due to lack of portal insulin and delayed pharmacokinetics of subcutaneous bolus insulin.

ii) Hepatic glucose uptake will be higher in participants after bariatric surgery compared with matched health controls due to accelerated glucose absorption and earlier and higher peak portal glucose and insulin concentrations.

DETAILED DESCRIPTION:
The liver has a central role in maintaining glucose homeostasis. During periods following food intake the liver stores glucose whilst during fasting periods it produces and releases glucose into the circulation. These key regulatory features prevent hyperglycaemia after meals via increase in hepatic glucose uptake and prevent hypoglycaemia during food deprivation via hepatic glucose output. Although the exact numbers are unknown, it is suggested that approximately 25%-30% of an oral glucose load are taken up by the liver. Since hepatic glucose uptake is closely linked with hepatic glycogen synthesis, the fraction of an oral glucose load that is converted to glycogen is similar or somewhat less. Other pathways downstream of hepatic glucose uptake are the conversion to lactate, oxidation to carbon dioxide (CO2) or synthesis of fatty acids. Glycogenolysis and gluconeogenesis contribute to hepatic glucose output, in yet unknown proportions. Key regulators of hepatic glucose metabolism act through diverse mechanisms. Hepatic glucose uptake is mainly regulated by the level of insulin, the rate of glucose appearance in the portal vein, the portal-peripheral glucose and insulin gradient and neuronal signalling1. Hepatic glucose production is regulated by the provision of substrates such as lactate and glycerol, allosteric control by metabolites such as glucose, and balance of hormones such as insulin, glucagon and catecholamines. An imbalance between hepatic glucose uptake and hepatic glucose output results in dysglycaemia which can be both hyper- or hypoglycaemia.

Hepatic glucose metabolism is dysregulated in a broad spectrum of diseases. Prime examples are type 1 and type 2 diabetes in which altered hepatic glucose handling contributes to hyperglycaemia, although via distinct mechanisms. Whereas in type 2 diabetes, insulin resistance and hence impaired suppression of hepatic glucose output is the key pathophysiological feature, lack of the portal-peripheral insulin gradient (insulin levels normally threefold higher in portal vein than in arterial blood due to drainage of secreted endogenous insulin into the portal vein) seems to be more relevant in type 1 diabetes. In the latter case absolute insulin deficiency and hence coverage of total insulin requirements by the exogenous subcutaneous route generates a very different vascular insulin profile compared with endogenously secreted insulin. Experiments in conscious dogs showed that glucose uptake is equally divided between the liver and muscle when insulin is infused via the portal vein, but when insulin is delivered peripherally the percentage of glucose taken up by the liver is less than half of normal. These findings suggest that peripherally delivered insulin cannot replicate the physiologic regulation of postprandial hepatic glucose uptake, but direct evidence in humans is currently lacking.

Another condition that is characterised by an altered portal milieu are patients having undergone bariatric surgery. The re-arrangement of the gastrointestinal tract substantially alters the portal milieu by accelerated glucose fluxes and higher and earlier gut peptide hormone patterns. The two most commonly performed bariatric surgery procedures, namely Roux-en-Y gastric bypass, which re-routes the small intestine to a small stomach pouch, and sleeve gastrectomy, which reduces the stomach to about 15% of its original size, significantly accelerate glucose absorption. It was recently demonstrated that this effects is more pronounced after Roux-en-Y-gastric bypass than sleeve gastrectomy. Accelerated glucose absorption leads to higher glucose concentrations in the portal vein. Of note, animal experiments using portal vein catheterization showed that under elevated glucose levels in the portal vein promote hepatic glucose uptake, however direct evidence in post-bariatric surgery patients is lacking.

Organ-specific substrate exchanges (uptake and output) can be best studied by measuring arterio-venous substrate concentration difference and organ blood supply. The additional use of isotopically labelled substrates further allows calculating intra-organ turnover rate. Although invasive, this method can be applied for most organs or tissue, such as the kidney, heart, brain or whole limbs. The liver's anatomical location and connection to the portal circulation makes the the calculation of arterio-venous-substrate gradient in humans particularly challenging, however. Surgical catheterization of the portal vein in humans is not possible for practical and ethical reasons. As a consequence, current non-invasive approaches in humans rely on the use of stable isotopes and can only provide an estimate of splanchnic glucose uptake (sum of liver and intestinal glucose utilisation) but do not allow for the quantification of hepatic glucose uptake.

Since it is generally assumed that the liver is the sole source of glucose production (an assumption essentially verified in normal condition, since the kidney appears to contribute less than 10% total glucose output), a simplified tracer approach with analysis of the systemic dilution of infused labelled glucose can reliably estimate hepatic (endogenous) glucose output. However, such isotope dilution cannot estimate hepatic glucose uptake, which has essentially been indirectly assessed in multiple (oral+iv) glucose tracers experiment and calculation of the systemic appearance of ingested labelled glucose. These measurements are however tightly dependent on the mathematical model used and hence remain semiquantitative. Furthermore, they do not allow to differentiate gut and hepatic glucose uptake.

Thus, the only way to directly assess hepatic glucose uptake is through highly invasive portal vein catheterization which requires animal models. Such models can simulate postprandial hepatic glucose handling but applicability to humans are limited. Current concepts of hepatic glucose uptake under different conditions mainly stem from animal experiments in which overnight fasted conscious dogs underwent portal vein catheterization.

From the above mentioned dilemma it follows that obtaining quantitative data on hepatic glucose uptake in humans requires a non-invasive approach such as imaging. Positron emission tomography (PET) scanning with the tracer fluorine-18 (F-18) fluorodeoxyglucose (FDG), called FDG-PET enables direct observation of tissue glucose uptake by quantifying radioactivity over time in vivo. Some researchers have thus suggested to use FDG-PET to study human glucose metabolism. However, FDG-PET confers the major downside of exposing individuals to remarkable amounts of radiation, a risk that is not considered justified for research purposes only. In addition FDG-PET does not inform on metabolism downstream of glucose uptake and the intravenous administration route of the radioactive glucose is not reflective of normal physiology.

Clearly, there is a demand for a non-invasive, non-radioactive and easily applicable approach to investigate human hepatic glucose metabolism including the quantification of hepatic glucose uptake. Deuterium metabolic imaging is a novel, non-invasive imaging approach that combines deuterium magnetic resonance spectroscopic imaging with oral intake or intravenous infusion of nonradioactive 2H-labeled substrates to generate three-dimensional metabolic maps. Deuterium metabolic imaging can reveal glucose metabolism beyond mere uptake and can be used with other Deuterium (2H)-labeled substrates as well. It has recently been demonstrated by De Feyter et al. that deuterium metabolic imaging allows mapping of glucose metabolism in the brain and liver of animal models and human subjects using 6,6-2H2-glucose. Deuterium metabolic imaging is a promising, non-invasive and easy-to-implement imaging technique that opens new avenues to address important knowledge gaps such as the extent and dynamics of postprandial hepatic glucose uptake and utilisation.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years
* Capacity to give informed consent
* Willingness to adhere to the study protocol

In group II (type 1 diabetes), the following criteria must be met in addition:

* T1D for ≥2 years or evidence of undetectable C-peptide (<100pmol/l with concomitant plasma glucose≥4.0mmol/l)
* HbA1c≤8.0mmol/l (64mmol/mol)

In group III (bariatric surgery), the following criteria must be met in addition:

* Female
* Bariatric surgery (Roux-en-Y gastric bypass or sleeve gastrectomy) ≥1 year ago
* Lack of a history of diabetes or pre-diabetes (HbA1c≤5.6% in the absence of anaemia)

Exclusion Criteria:

* Pregnancy, planned pregnancy or breastfeeding
* Medication that interfere with glucose metabolism (participation requires discontinuation of these agents at least one week before the study visit) except for individuals with type 1 diabetes
* History of gastrointestinal surgery (other than bariatric surgery for group III)
* Known kidney, liver or heart disease
* Claustrophobia
* Contraindications to magnetic resonance imaging according to designated questionnaire
* Substance abuse
* Physical or psychological condition likely to interfere with the normal conduct of the study and interpretation of the study results as judged by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy participants will be recruited through advertisement on the hospital staff website and website of the Medical faculty according to Swissethics guidelines. Patients with type 1 diabetes and post-bariatric surgery patients will be recruited through referring physicians from the University Hospital Bern or colleagues from local private outpatient clinics.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2022-04-21 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Intrahepatic free glucose concentration | Over postprandial period (0 to 150 minutes post glucose-ingestion)

SECONDARY OUTCOMES:
Postprandial hepatic glycogen increment | Over postprandial period (0 to 150 minutes post glucose-ingestion)
Postprandial glucose exposure | Over postprandial period (0 to 150 minutes post glucose-ingestion)
  Incremental area under the glucose concentration curve
Postprandial glucagon exposure | Over postprandial period (0 to150 minutes post glucose-ingestion)
  Incremental area under the glucagon concentration curve
Postprandial insulin secretion | Over postprandial period (0 to 150 minutes post glucose-ingestion)
  Calculated using the Oral Glucose minimal Model
Postprandial insulin exposure | Over postprandial period (0 to 150 minutes post glucose-ingestion)
  Incremental area under the insulin concentration curve
Postprandial insulin clearance | Over postprandial period (0 to 150 minutes post glucose-ingestion)
Postprandial whole body insulin sensitivity | Over postprandial period (0 to 150 minutes post glucose-ingestion)
  Calculated using the Oral Glucose Minimal Model
Postprandial hepatic glucose production | Over postprandial period (0 to 150 minutes post glucose-ingestion)
  Estimated using the single tracer oral minimal model based on the ingested dose of 6,6-2H2-glucose and plasma 6,6-2H2-glucose enrichment
First-pass hepatic extraction of glucose | Over postprandial period (0 to 150 minutes post glucose-ingestion)

OTHER OUTCOMES:
Quantification of 2H-labelled metabolites other than glucose (i.e. lactate, glutamate/glutamine, water) | Over postprandial period (0 to 150 minutes post glucose-ingestion)
Changes in intrahepatocellular lipid (IHCL) | Over postprandial period (0 to 150 minutes post glucose-ingestion)

CONTACTS AND LOCATIONS:
Overall Officials: Lia Bally, MD, PhD, Principal Investigator — University Hospital Bern & University of Bern
Locations (1):
- Inselspital, Bern University Hospital and University Hospital of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No